CLINICAL TRIAL: NCT02165501
Title: Jena Sepsis Registry - a Sepsis-registry for Long Term Outcomes
Brief Title: Jena Sepsis Registry
Acronym: JenaSepsisReg
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, Jochen Gensichen, MD, MA, MPH, Professor and Chair, Jena University Hospital
Other Study IDs: 3218-08/11; FZ 01 E0 1002 (Other Grant/Funding Number: Federal Ministry of Education and Research (BMBF))
Record Dates: First submitted 2014-06-11; First posted 2014-06-17 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Severe Sepsis or Septic Shock (ICD-10-GM, R65.0, R65.1)
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Despite the burden of severe sepsis and septic shock deficiencies in the quality of sepsis management are recognized. Investigators present a population-based registry with easy feasibility as part of German Center for Sepsis Control & Care (CSCC). All ICU patients of the Jena University Hospital, Germany will be screened for inclusion (severe sepsis or septic shock). Baseline data on ICU- and hospital care will be extracted from patient records at ICU discharge. The primary outcome is change in all-cause mortality from baseline to follow up at 6, 12, 24, 36, 48 and 60 months after diagnosis of sepsis. Follow-up data will be collected from the primary care provider of the patient. The registry may provide valid data on quality in sepsis care.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated in one of the ICUs will be enrolled if they were 18 years or older and fulfill the diagnostic criteria of severe sepsis or septic shock (ICD-10-GM, R65.0, R65.1) (19), (20).
* Diagnosis of severe sepsis or septic shock requires the following criteria: a microbiologically documented and/or clinically evident infection, at least two of the four criteria of the systemic inflammatory response syndrome (SIRS) and at least one new organ dysfunction, remote from the site of infection.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients will be selected from Jena University Hospital, Germany
Sampling Method: Non-Probability Sample
Enrollment: 1995 (Actual)
Dates: Start 2011-01; Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | change from baseline to 6,12, 24, 36, 48 and 60 months after ICU discharge
  based on data from hospital records as well as patient records of the primary care provider.

CONTACTS AND LOCATIONS:
Locations (1):
- Jena University Hospital, Jena, Germany

REFERENCES:
- See also: Related Info — http://www.allgemeinmedizin.uni-jena.de